## INFORMED CONSENT FORM

**Study Title:** The Effect of Positive Psychotherapy-Based Self-Compassion Training on Internalized Stigma, Loneliness, and Empathy Levels of Parents of Children With Special Needs

NCT Number: NCTXXXXXXXX Document Date: August 1, 2025

#### **Informed Consent Statement**

This study has received written approval from the Institutional Review Board of Batman University Non-Interventional Clinical Research Ethics Committee. We invite you to voluntarily participate in this research.

Participation is completely optional, and you have the right to withdraw at any time without any consequences.

### **Purpose of the Study**

This study aims to investigate the effects of positive psychotherapy-based self-compassion training on internalized stigma, loneliness, and empathy levels among parents of children with special needs.

## **What Participation Involves**

If you agree to participate:

- You will be asked to attend and engage in positive psychotherapy-based selfcompassion training sessions for a specified period.
- You will complete questionnaires measuring internalized stigma, loneliness, and empathy levels.

#### **Risks and Benefits**

During the study, you may experience emotional reactions while reflecting on your caregiving experience and feelings. If you feel any discomfort, you may stop at any time.

## **Confidentiality**

All information will be kept confidential and will only be used for research purposes.

# **Voluntary Participation**

You may refuse to participate or withdraw at any time without providing a reason or facing any negative consequences.

If you agree to participate, please sign below. You will receive a copy of this form.

| Participant Information and Consent | |
|-------------------------------------|---------------|
| Participant's Full Name: | |
| Address: | |
| Phone Number: | |
| Signature: | Date://2025 |
| Researcher Information | |
| Researcher's Full Name and Title: | |
| Institution / Address: | |
| Phone Number: | |
| Signature: | Date: / /2025 |